CLINICAL TRIAL: NCT01258387
Title: A Phase 1, Double-Blind, Placebo-Controlled Study of Single Ascending Doses of GGF2 in Patients With Left Ventricular Dysfunction and Symptomatic Heart Failure
Brief Title: Single Ascending Doses of GGF2 in Patients With Left Ventricular Dysfunction and Symptomatic Heart Failure
Acronym: GGF2-1101-1
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Acorda Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 1101.1
Record Dates: First submitted 2010-12-08; First posted 2010-12-13 (Estimated); Results first posted 2014-07-01 (Estimated); Last update posted 2014-07-01 (Estimated); Status verified 2014-06

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — Neuregulins

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- GGF2 (Placebo Comparator): Seven dosing cohorts: 2 patients randomized to receive 1 GGF2, 1 placebo; if no drug-related dose-limiting toxicities in GGF2-treated patient, other 4 patients in cohort will be randomized (3:1) and dosed
  Interventions: Drug: Glial growth factor 2/ Neuregulin 1β3; Other: Placebo

INTERVENTIONS:
Drug: Glial growth factor 2/ Neuregulin 1β3
  Other Names: Recombinant Human Glial Growth Factor 2
Other: Placebo

SUMMARY:
Study to determine the safety, tolerability, pharmacokinetics and immunogenicity of single intravenous administrations of GGF2 in patients with heart failure.

DETAILED DESCRIPTION:
Phase 1, double-blind, placebo-controlled, dose escalation study to determine the safety, tolerability, pharmacokinetics and immunogenicity of single intravenous administrations of GGF2 in cohorts of patients with left ventricular dysfunction and symptomatic heart failure.

ELIGIBILITY:
Inclusion Criteria:

1. Left ventricular ejection fraction (LVEF) between 10% and 40%.
2. Male or female, aged 18 to 75 years, inclusive.

Exclusion Criteria:

1. Received any investigational agent or participation in any clinical study of an investigational agent or investigational therapy up to 30 days prior to the screening visit.
2. Use of any new prescription medication up to 14 days prior to receiving investigational drug.
3. Patients with known specific hepatic disease; bilirubin >2 mg/dL, SGOT > 100 IU.
4. Patients with a history of hepatic impairment (hepatitis B and C).
5. Serum creatinine >2.5 mg/dL.
6. Documented stroke or transient ischemic attack (TIA) within 60 days of study enrollment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2010-12; Primary Completion 2012-12 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Caggiano, MD, PhD, Study Director — Acorda Therapeutics
Locations (2):
- United States (2):
  - The Medical Group of Saint Joseph's, Atlanta, Georgia
  - Vanderbilt University, Nashville, Tennessee

RESULTS

PARTICIPANT FLOW:
Recruitment Details: After informed consent, 40 patients with symptomatic Heart Failure (HF) were randomized (4:2) to GGF2 or placebo in 7 ascending dose cohorts. Patients were observed in hospital for 30 hours, then evaluated for adverse effects at 1, 2, 4, 12, and 24 weeks after infusion.
Pre-assignment Details: There were six patients in each cohort/dose level, four received active treatment (GGF2) and two received placebo. In each dose level, the first two patients were randomized 1:1 to GGF2 or placebo and monitored for safety prior to randomizing the remaining patients in the cohort 3:1. GGF2 or placebo was administered as an IV infusion.
Groups:
- GGF2 First Dose: First dosing: 1 GGF2, 1 pbo; if no drug-related dose-limiting toxicities in GGF2-treated patient, other 4 patients in cohort randomized (3:1) and dosed
- GGF2 Second Escalated Dose: Second dosing: 1 GGF2, 1 pbo; if no drug-related dose-limiting toxicities in GGF2-treated patient, other 4 patients in cohort randomized (3:1) and dosed
- GGF2 Third Escalated Dose: Third dosing: 1 GGF2, 1 pbo; if no drug-related dose-limiting toxicities in GGF2-treated patient, other 4 patients in cohort randomized (3:1) and dosed
- GGF2 Fourth Escalated Dose: Fourth dosing: 1 GGF2, 1 pbo; if no drug-related dose-limiting toxicities in GGF2-treated patient, other 4 patients in cohort randomized (3:1) and dosed
- GGF2 Fifth Escalated Dose: Fifth dosing: 1 GGF2, 1 pbo; if no drug-related dose-limiting toxicities in GGF2-treated patient, other 4 patients in cohort randomized (3:1) and dosed
- GGF2 Sixth Escalated Dose: Sixth dosing: 1 GGF2, 1 pbo; if no drug-related dose-limiting toxicities in GGF2-treated patient, other 4 patients in cohort randomized (3:1) and dosed .
- GGF2 Seventh Escalataed Dose: Seventh dosing: 1 GGF2, 1 pbo; if no drug-related dose-limiting toxicities in GGF2-treated patient, other 4 patients in cohort randomized (3:1) and dosed
Period: Overall Study
Arm/Group | GGF2 First Dose | GGF2 Second Escalated Dose | GGF2 Third Escalated Dose | GGF2 Fourth Escalated Dose | GGF2 Fifth Escalated Dose | GGF2 Sixth Escalated Dose | GGF2 Seventh Escalataed Dose
Started | 6 | 6 | 6 | 6 | 6 | 6 | 4
Patients Randomized to GGF2 | 4 | 4 | 4 | 4 | 4 | 4 | 3
Patients Randomized to Placebo | 2 | 2 | 2 | 2 | 2 | 2 | 1
Completed | 6 | 6 | 6 | 6 | 6 | 6 | 4
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety Population. Consists of all patients who took one of the double-blind investigational drugs.
Groups:
- Placebo: Patients in each of 7 cohorts randomized to Placebo
- GGF2 First Dose: First dosing: patients in cohort randomized to GGF2
- GGF2 Second Escalated Dose: Second dosing: patients in cohort randomized to GGF2
- GGF2 Third Escalated Dose: Third dosing: patients in cohort randomized to GGF2
- GGF2 Fourth Escalated Dose: Fourth dosing: patients in cohort randomized to GGF2
- GGF2 Fifth Escalated Dose: Fifth dosing: patients in cohort randomized to GGF2
- GGF2 Sixth Escalated Dose: Sixth dosing: patients in cohort randomized to GGF2.
- GGF2 Seventh Escalataed Dose: Seventh dosing: patients in cohort randomized to GGF2
- Total: Total of all reporting groups
Arm/Group | Placebo | GGF2 First Dose | GGF2 Second Escalated Dose | GGF2 Third Escalated Dose | GGF2 Fourth Escalated Dose | GGF2 Fifth Escalated Dose | GGF2 Sixth Escalated Dose | GGF2 Seventh Escalataed Dose | Total
Number analyzed (Participants) | 13 | 4 | 4 | 4 | 4 | 4 | 4 | 3 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.7 (13.21) | 52.0 (5.72) | 58.5 (7.59) | 56.8 (10.05) | 65.3 (5.85) | 58.5 (8.85) | 59.0 (4.97) | 61.0 (9.17) | 57.4 (9.83)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 0 | 2 | 1 | 1 | 0 | 0 | 7
  Male | 12 | 2 | 4 | 2 | 3 | 3 | 4 | 3 | 33
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 13 | 4 | 4 | 4 | 4 | 4 | 4 | 3 | 40
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Safety of Single Ascending Doses of GGF2 Via an Assessment of the Toxicology Profile as Measured by Treatment Emergent Adverse Events (TEAEs)
Description: Safety/ tolerability of single dose; cumulative safety over 6 months
  TEAEs are defined as adverse events with date of onset (or worsening) on or after the start date of double-blind treatment and no more than 28 days from the start date of double-blind treatment.
Time Frame: 6 months
Population: Safety population
Measure: Number; unit: participants
Arm/Group | Placebo | GGF2 First Dose | GGF2 Second Escalated Dose | GGF2 Third Escalated Dose | GGF2 Fourth Escalated Dose | GGF2 Fifth Escalated Dose | GGF2 Sixth Escalated Dose | GGF2 Seventh Escalataed Dose
Number analyzed (Participants) | 13 | 4 | 4 | 4 | 4 | 4 | 4 | 3
participants
  Having Any TEAEs - Yes | 6 | 4 | 4 | 2 | 4 | 4 | 4 | 3
  Having Any TEAEs - No | 7 | 0 | 0 | 2 | 0 | 0 | 0 | 0
  Having TEAEs Maximum Severity Mild | 5 | 1 | 3 | 0 | 1 | 1 | 2 | 0
  Having TEAEs Maximum Severity Moderate | 1 | 3 | 1 | 2 | 2 | 1 | 2 | 2
  Having TEAEs Maximum Severity Severe | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 1
  Having TEAEs Maximum Toxicity Grade Mild | 5 | 1 | 3 | 0 | 1 | 1 | 2 | 1
  Having TEAEs Maximum Toxicity Grade Moderate | 0 | 3 | 1 | 2 | 2 | 1 | 2 | 1
  Having TEAEs Maximum Toxicity Grade Severe | 1 | 0 | 0 | 0 | 1 | 2 | 0 | 1
  TEAEs Maximum Toxicity Grade Life-Threatening | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Having TEAEs Maximum Toxicity Grade Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Relationship to Study Drug -Not Related | 5 | 1 | 1 | 1 | 3 | 1 | 1 | 0
  Relationship to Study Drug -Related | 1 | 3 | 3 | 1 | 1 | 3 | 3 | 3
  Withdrew Due to TEAEs - Yes | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Withdrew Due to TEAEs - NO | 13 | 4 | 4 | 4 | 4 | 4 | 4 | 3

2. Secondary Outcome: Change From Baseline of Two-Dimensional Echocardiogram (2D-ECHO) Measured by Ejection Fraction (EF)
Description: An echocardiogram is a type of ultrasound test that uses high-pitched sound waves that are sent through a device called a transducer. The device picks up echoes of the sound waves as they bounce off the different parts of your heart. These echoes are turned into moving pictures of your heart that can be seen on a video screen.¹
  Ejection fraction is a measurement of the percentage of blood leaving your heart each time it contracts.²
  ¹http://wakeinternalmedicine.com/services-and-procedures/services/radiology/2d-echo/
  ²http://www.mayoclinic.org/ejection-fraction/expert-answers/faq-20058286
Time Frame: Screening, day 8, day 14, day 28, and 3 months post-dose
Population: Safety Population
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Placebo | GGF2 First Dose | GGF2 Second Escalated Dose | GGF2 Third Escalated Dose | GGF2 Fourth Escalated Dose | GGF2 Fifth Escalated Dose | GGF2 Sixth Escalated Dose | GGF2 Seventh Escalataed Dose
Number analyzed (Participants) | 13 | 4 | 4 | 4 | 4 | 4 | 4 | 3
percent change
  Day 8 | -0.82 (6.582) | 4.75 (8.180) | 5.00 (7.528) | 2.50 (5.196) | 4.25 (4.272) | -1.25 (4.992) | 5.33 (8.083) | 4.33 (3.055)
  Day 14 | -1.12 (7.880) | -5.00 (7.257) | 5.00 (10.863) | 2.00 (4.546) | 4.23 (8.328) | 2.13 (5.360) | 11.55 (10.007) | 7.10 (8.627)
  Day 28 | -0.27 (8.584) | -2.00 (9.345) | 8.50 (10.472) | 4.00 (2.449) | 8.00 (2.000) | 5.75 (2.500) | 12.00 (5.099) | 10.00 (7.550)
  3 Months | 1.88 (8.588) | -3.75 (6.397) | 0.78 (8.418) | 0.75 (4.031) | 7.25 (8.770) | 4.50 (7.724) | 9.00 (5.598) | 15.00 (13.000)

3. Secondary Outcome: Change From Baseline of 2D-ECHO Measured by End-Diastolic Volume (EDV)
Description: EDV is the amount of blood in the ventricle immediately before a cardiac contraction begins; used as a measurement of diastolic function.¹
  ¹http://medical-dictionary.thefreedictionary.com/end-diastolic+volume
Time Frame: Screening, day 8, day 14, day 28, and 3 months post-dose
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Milliliter(s)
Arm/Group | Placebo | GGF2 First Dose | GGF2 Second Escalated Dose | GGF2 Third Escalated Dose | GGF2 Fourth Escalated Dose | GGF2 Fifth Escalated Dose | GGF2 Sixth Escalated Dose | GGF2 Seventh Escalataed Dose
Number analyzed (Participants) | 13 | 4 | 4 | 4 | 4 | 4 | 4 | 3
Milliliter(s)
  Day 8 | -14.89 (74.125) | 27.50 (27.538) | 1.98 (29.028) | -10.60 (59.288) | -2.15 (11.098) | -35.00 (36.341) | 17.00 (23.763) | 7.33 (5.859)
  Day 14 | -41.59 (55.252) | 31.95 (9.450) | -10.25 (56.119) | -32.83 (44.543) | -22.25 (30.609) | -26.50 (33.071) | -23.50 (61.474) | 17.85 (19.587)
  Day 28 | -25.85 (63.405) | 13.60 (21.750) | 49.18 (52.333) | -21.05 (41.282) | 10.50 (54.482) | -15.80 (20.785) | -15.25 (74.384) | -3.30 (13.262)
  3 Months | -25.72 (109.056) | 2.85 (43.507) | -8.00 (46.168) | 48.78 (66.896) | -20.00 (36.615) | -39.85 (52.616) | -12.98 (116.297) | 4.07 (30.624)

4. Secondary Outcome: Change From Baseline of 2D-ECHO Measured by End-Systolic Volume (ESV)
Description: ESV is the volume of blood remaining in each ventricle at the end of systole.¹
  ¹http://medical-dictionary.thefreedictionary.com/end-diastolic+volume
Time Frame: Screening, day 8, day 14, day 28, and 3 months post-dose
Population: Safety Population
Measure: Mean (Standard Deviation); unit: Milliliter(s)
Arm/Group | Placebo | GGF2 First Dose | GGF2 Second Escalated Dose | GGF2 Third Escalated Dose | GGF2 Fourth Escalated Dose | GGF2 Fifth Escalated Dose | GGF2 Sixth Escalated Dose | GGF2 Seventh Escalataed Dose
Number analyzed (Participants) | 13 | 4 | 4 | 4 | 4 | 4 | 4 | 3
Milliliter(s)
  Day 8 | -0.92 (79.285) | 12.38 (31.669) | -6.98 (29.443) | -15.95 (44.215) | -5.25 (15.392) | -26.50 (30.490) | -9.00 (29.017) | -3.23 (12.894)
  Day 14 | -19.08 (76.181) | 33.20 (14.200) | -14.40 (30.961) | -27.65 (31.115) | -15.00 (20.314) | -27.25 (39.339) | -31.75 (58.750) | 4.10 (2.970)
  Day 28 | -3.48 (92.552) | 10.88 (22.885) | 22.05 (41.977) | -23.45 (30.330) | -8.88 (25.873) | -24.75 (26.725) | -28.75 (60.808) | -16.30 (8.311)
  3 Months | -12.65 (128.433) | 6.30 (32.395) | -0.45 (32.211) | 27.80 (43.414) | -21.25 (23.782) | -39.08 (48.393) | -18.58 (87.663) | -10.73 (36.960)

ADVERSE EVENTS:
Time Frame: 6 months
Description: Serious Treatment Emergent Adverse Events (TEAE) are defined as serious Adverse Events (AE) with date of onset (or worsening) on or after the start date of double-blind treatment.
Groups:
- GGF2 First Dose: First dosing: 1 GGF2, 1 pbo; if no drug-related dose-limiting toxicities in GGF2-treated patient, other 4 patients in cohort will be randomized (3:1) and dosed
- GGF2 Second Escalated Dose: Second dosing: 1 GGF2, 1 pbo; if no drug-related dose-limiting toxicities in GGF2-treated patient, other 4 patients in cohort will be randomized (3:1) and dosed
- GGF2 Third Escalated Dose: Third dosing: 1 GGF2, 1 pbo; if no drug-related dose-limiting toxicities in GGF2-treated patient, other 4 patients in cohort will be randomized (3:1) and dosed
- GGF2 Fourth Escalated Dose: Fourth dosing: 1 GGF2, 1 pbo; if no drug-related dose-limiting toxicities in GGF2-treated patient, other 4 patients in cohort will be randomized (3:1) and dosed
- GGF2 Fifth Escalated Dose: Fifth dosing: 1 GGF2, 1 pbo; if no drug-related dose-limiting toxicities in GGF2-treated patient, other 4 patients in cohort will be randomized (3:1) and dosed
- GGF2 Sixth Escalated Dose: Sixth dosing: 1 GGF2, 1 pbo; if no drug-related dose-limiting toxicities in GGF2-treated patient, other 4 patients in cohort will be randomized (3:1) and dosed .
- GGF2 Seventh Escalataed Dose: Seventh dosing: 1 GGF2, 1 pbo; if no drug-related dose-limiting toxicities in GGF2-treated patient, other 4 patients in cohort will be randomized (3:1) and dosed
Arm/Group | Placebo | GGF2 First Dose | GGF2 Second Escalated Dose | GGF2 Third Escalated Dose | GGF2 Fourth Escalated Dose | GGF2 Fifth Escalated Dose | GGF2 Sixth Escalated Dose | GGF2 Seventh Escalataed Dose
Serious Adverse Events (participants affected / at risk) | 0/13 | 1/4 | 1/4 | 0/4 | 1/4 | 0/4 | 0/4 | 1/3
Other Adverse Events (participants affected / at risk) | 6/13 | 4/4 | 4/4 | 2/4 | 4/4 | 4/4 | 4/4 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=13) | GGF2 First Dose (N=4) | GGF2 Second Escalated Dose (N=4) | GGF2 Third Escalated Dose (N=4) | GGF2 Fourth Escalated Dose (N=4) | GGF2 Fifth Escalated Dose (N=4) | GGF2 Sixth Escalated Dose (N=4) | GGF2 Seventh Escalataed Dose (N=3)
Angina pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hy's law case (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Viral infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=13) | GGF2 First Dose (N=4) | GGF2 Second Escalated Dose (N=4) | GGF2 Third Escalated Dose (N=4) | GGF2 Fourth Escalated Dose (N=4) | GGF2 Fifth Escalated Dose (N=4) | GGF2 Sixth Escalated Dose (N=4) | GGF2 Seventh Escalataed Dose (N=3)
Headache (Nervous system disorders) | 0 (0) | 2 | 2 | 1 | 0 | 2 | 2 | 1
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lethargy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Sinus headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 2 | 0 | 0 | 1 | 1 | 2 | 1 | 2
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 2
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Abdominal Pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal tenderness (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Fatigue (General disorders) | 1 | 1 | 0 | 1 | 0 | 2 | 2 | 0
Feeling hot (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Infusion site pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Injection site haematoma (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Injection site scab (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pyrexia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Influenza like illness (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Brain natriuretic peptide increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Blood chloride increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Blood potassium increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Glomerular filtration rate decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Heart rate increased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Weight decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1 | 2 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0
Nasal conjestion (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1
Flushing (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Hot flush (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vein pain (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Viral infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Fluid retention (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Gout (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Angina pectoris (Cardiac disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Cardiac flutter (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Muscle strain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Chromaturia (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vitreous floaters (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hy's law case (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor (Acorda) has the right to review and comment on proposed publications within a specified time frame, up to 60 days; multi-center trials require joint publication unless specifically permitted otherwise.